CLINICAL TRIAL: NCT06678373
Title: Monitoring JE Antibody Levels in Healthy Populations and Immunization Strategy in Low-Prevalence Areas
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liaoning Chengda Biotechnology CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDB-JE-PM-2023004
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A(Ages 6 to 17) (Experimental): The patient needs to receive 1 dose of inactivated Japanese encephalitis vaccine.
  Interventions: Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine
- Group B(Ages 18 to 39) (Experimental): The patient needs to receive 2 doses of inactivated Japanese encephalitis vaccine, with an interval of 28 days.
  Interventions: Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine
- Group C(C1 Age 18-39 years) (Experimental): The patient needs to receive 2 doses of inactivated Japanese encephalitis vaccine, with an interval of 7 days.
  Interventions: Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine
- Group C(C2 Age 40-59 years) (Experimental): The patient needs to receive 2 doses of inactivated Japanese encephalitis vaccine, with an interval of 7 days.
  Interventions: Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine
- Group C(C3 Age 60 years and above) (Experimental): The patient needs to receive 2 doses of inactivated Japanese encephalitis vaccine, with an interval of 7 days.
  Interventions: Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine

INTERVENTIONS:
Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine — The patient needs to receive 1 dose of inactivated Japanese encephalitis vaccine.
  Arms: Group A(Ages 6 to 17)
Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine — The patient needs to receive 2 doses of inactivated Japanese encephalitis vaccine, with an interval of 28 days.
  Arms: Group B(Ages 18 to 39)
Biological: Liaoning Chengda Inactivated Japanese Encephalitis Vaccine — The patient needs to receive 2 doses of inactivated Japanese encephalitis vaccine, with an interval of 7 days.
  Arms: Group C(C1 Age 18-39 years); Group C(C2 Age 40-59 years); Group C(C3 Age 60 years and above)

SUMMARY:
This study aims to assess the neutralizing antibody levels and prevalence risk of Japanese encephalitis among residents in low-endemic areas, as well as to evaluate the immunogenicity, safety, and immune persistence of the inactivated Japanese encephalitis vaccine across different age groups in healthy populations. The study uses an open-label, single-arm trial design with a sample size of 250 participants. Primary endpoints include pre- and post-vaccination serum neutralizing antibody levels, seroconversion rates, and incidence of adverse events.

DETAILED DESCRIPTION:
This study aims to gain an in-depth understanding of neutralizing antibody levels against Japanese encephalitis among residents in low-endemic areas to assess potential outbreak risks and to evaluate the immunogenicity, safety, and immune persistence of the inactivated Japanese encephalitis vaccine across different age groups in a healthy population. This open-label, single-arm trial is structured in two phases: Phase I will involve stratified sampling of residents aged 6 years and older for serological testing, followed by administration of the inactivated JE vaccine to assess safety, with serological testing conducted 28 days post-vaccination. Phase II will conduct serological testing 365 days post-primary immunization to evaluate immune persistence.

The target population includes residents aged 6 and older, divided into Group A (ages 6-17), Group B (ages 18-39), and Group C (ages 18+), with different vaccine dosages for each group. Inclusion criteria encompass age, health status, and informed consent, while exclusion criteria cover allergies, serious illness, and recent vaccination. Primary endpoints will include pre- and post-vaccination serum neutralizing antibody levels, seroconversion rates, average antibody levels, and post-vaccination adverse event incidence. The project is scheduled to begin in October 2024 and conclude in December 2026, with the primary research unit being the Liaoning Provincial Center for Disease Control and Prevention, aiming to provide a scientific basis for JE control and prevention in this region.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents aged 6 years (inclusive) and older;
* Healthy individuals as determined clinically after inquiring about medical history and conducting relevant physical examinations;
* Individuals who meet the vaccination criteria for the inactivated Japanese encephalitis vaccine (Vero cells);
* Participants must provide informed consent to receive vaccination and blood c collection; minors must obtain informed consent from their guardians;
* Participants planned to be included in Group A must have previously completed the full vaccination schedule for the Japanese encephalitis vaccine (including live attenuated vaccine or inactivated vaccine).

Exclusion Criteria:

* Participants are unwilling to sign the informed consent form;
* History of allergy to the vaccine or its components, severe adverse reactions to the vaccine such as allergies, urticaria, breathing difficulties, angioedema, or abdominal pain;
* Individuals with encephalopathy, uncontrolled epilepsy, and other progressive neurological diseases;
* History of seizures or convulsions, or family history of psychiatric disorders;
* Presence of congenital malformations or developmental disorders, genetic defects, and severe malnutrition;
* Individuals with autoimmune diseases, congenital or acquired immunodeficiencies, or family history of autoimmune diseases or immunodeficiencies;
* Any acute diseases or acute exacerbations of chronic diseases in the past 7 days;
* Treatment with immunosuppressants, anti-allergy treatments, cytotoxic therapies, or inhaled corticosteroids (excluding corticosteroid spray treatments for allergic rhinitis or topical corticosteroid treatments for acute non-complicated dermatitis) in the past 6 months;
* Administration of immunoglobulin injections within 1 month prior to vaccination;
* Individuals with fever before vaccination, with axillary temperature >37.0°C;
* History of Japanese encephalitis;
* Other factors deemed inappropriate for participation in the clinical observational study as determined by the researcher;
* Participants planned for inclusion in Groups B and C must have received the Japanese encephalitis vaccine (including live attenuated vaccine and inactivated vaccine) in the past;
* Pregnant women.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of JE neutralizing antibody levels in low-prevalence areas to evaluate the risk of JE transmission. | Prior to administration of the first vaccine dose.
  Before administering the first dose of the vaccine, at least 3 ml of the recipient's venous blood will be collected. Transport the serum under frozen conditions to the testing laboratory for analysis. The serum Japanese encephalitis neutralizing antibodies will be detected using the Plaque Reduction Neutralization Test (PRNT50). A neutralizing antibody titer of < 1:10 before vaccination is considered negative, while a titer of ≥ 1:10 after vaccination is considered positive. If the pre-vaccination antibody titer is ≥ 1:10, an increase of fourfold or more in the post-vaccination antibody titer is also considered a positive result.
Seroconversion rate and average neutralizing antibody levels against JE on the 28th day after vaccination. | On the 28th day after vaccination.
  After completing all doses of the trial, collect at least 3 ml of venous blood from the subjects on day 28. Transport the serum under frozen conditions to the testing laboratory for analysis. The serum Japanese encephalitis neutralizing antibodies will be detected using the Plaque Reduction Neutralization Test (PRNT50). A neutralizing antibody titer of < 1:10 before vaccination is considered negative, while a titer of ≥ 1:10 after vaccination is considered positive. If the pre-vaccination antibody titer is ≥ 1:10, an increase of fourfold or more in the post-vaccination antibody titer is also considered a positive result.

SECONDARY OUTCOMES:
Seroconversion rate and average neutralizing antibody levels against JE on the 365th day after vaccination. | On the 365th day after vaccination.
  After completing all doses of the trial, collect at least 3 ml of venous blood from the subjects on day 365. Transport the serum under frozen conditions to the testing laboratory for analysis. The serum Japanese encephalitis neutralizing antibodies will be detected using the Plaque Reduction Neutralization Test (PRNT50). A neutralizing antibody titer of < 1:10 before vaccination is considered negative, while a titer of ≥ 1:10 after vaccination is considered positive. If the pre-vaccination antibody titer is ≥ 1:10, an increase of fourfold or more in the post-vaccination antibody titer is also considered a positive result.
Adverse event rate | Within 30 days after vaccination.
  1. The incidence, severity, and correlation of any adverse events (AEs) at the injection site (local) and non-injection site (systemic) within 30 minutes after each dose;
  2. The incidence, severity, and correlation of AEs within 0-7 days after each dose;
  3. The incidence and correlation of all AEs and serious adverse events (SAEs) occurring within 30 days after the complete vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Fang, Principal Investigator — Liaoning Provincial Center for Disease Control and Prevention
Locations (1):
- Liaoning Provincial Center for Disease Control and Prevention, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No